CLINICAL TRIAL: NCT06105151
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Food Effects of a Single Oral VV119 Capsule in Healthy Chinese Volunteers
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics and Food Effects of VV119 Capsules in Chinese Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VV119-01
Record Dates: First submitted 2023-10-17; First posted 2023-10-27 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part Ⅰ - Single Ascending Dose (SAD) study: Experimental (Experimental): Subjects will receive VV119 orally for single dose.
  Interventions: Drug: VV119(SAD)
- Part Ⅰ - Single Ascending Dose (SAD) study: Placebo (Experimental): Subjects will receive VV119 placebo orally for single dose.
  Interventions: Drug: VV119 Placebo(SAD)
- Part Ⅱ - Food Effect (FE) study: Experimental (Experimental): Subjects will receive VV119 orally for single dose.
  Interventions: Drug: VV119(FE)

INTERVENTIONS:
Drug: VV119(SAD) — VV119 0.2 mg Group: 2 subjects will receive VV119 0.2 mg, orally; VV119 0.5 mg Group: 6 subjects will receive VV119 0.5 mg, orally; VV119 1 mg Group: 6 subjects will receive VV119 1 mg, orally; VV119 2 mg Group: 6 subjects will receive VV119 2 mg, orally; VV119 3 mg Group:6 subjects will receive VV119 3 mg, orally; VV119 4.5 mg Group:6 subjects will receive VV119 4.5 mg, orally; VV119 6 mg Group:6 subjects will receive VV119 6 mg, orally; VV119 8 mg Group:6 subjects will receive VV119 8 mg, orally; VV119 10 mg Group:6 subjects will receive VV119 10 mg, orally;
  Arms: Part Ⅰ - Single Ascending Dose (SAD) study: Experimental
Drug: VV119 Placebo(SAD) — VV119 0.5 mg Group: 2 subjects will receive VV119 Placebo 0.5 mg, orally; VV119 1 mg Group: 2 subjects will receive VV119 Placebo 1 mg, orally; VV119 2 mg Group: 2 subjects will receive VV119 Placebo 2 mg, orally; VV119 3 mg Group:2 subjects will receive VV119 Placebo 3 mg, orally; VV119 4.5 mg Group:2 subjects will receive VV119 Placebo 4.5 mg, orally; VV119 6 mg Group:2 subjects will receive VV119 Placebo 6 mg, orally; VV119 8 mg Group:2 subjects will receive VV119 Placebo 8 mg, orally; VV119 10 mg Group:2 subjects will receive VV119 Placebo 10 mg, orally;
  Arms: Part Ⅰ - Single Ascending Dose (SAD) study: Placebo
Drug: VV119(FE) — A：2 mg VV119, following an overnight fast of at least 10 hours for Period 1; 2mg VV119, administered 30 minutes after the start of a high-fat meal for Period 2; B: 2mg VV119, administered 30 minutes after the start of a high-fat meal for Period 1;2mg VV119, following an overnight fast of at least 10 hours for Period 2；
  Arms: Part Ⅱ - Food Effect (FE) study: Experimental

SUMMARY:
This study will consist of 2 parts: Part Ⅰ - Single Ascending Dose (SAD) study, Part Ⅱ - Food Effect (FE) study

DETAILED DESCRIPTION:
Part Ⅰ were designed as single-center, randomized, double-blind, placebo-controlled, dose-escalation trials to assess the safety, tolerability, pharmacokinetic (PK) of single oral doses of VV119 in healthy adult subjects.

Part Ⅱ is a single-center, randomized, open label, 2×2 crossover design to assess the high-fat meal effects on PK of a single oral dose of VV119 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males:aged 18 to 45 years old, males ,Body weight no less than 50.0 kg ; females :Aged 18 to 60 years old ,Body weight no less than 45.0 kg ,Body Mass Index of 19.0 to 26.0kg/m2,
2. Medically healthy, Physical examination, vital signs examination, laboratory examination, electrocardiogram examination results were normal or abnormal without clinical significance,
3. Males subjects who are willing to take effective contraceptive during the study and within 3 months after the study completed; females not of child-bearing potential,
4. Subjects who are able to understand and follow study plans and instructions; Subjects who have voluntarily decided to participate in this study, and signed the informed consent form.

Exclusion Criteria:

Unless otherwise noted, the exclusion criteria were consistent for subjects in the SAD study and FE study. The following subjects will be excluded:

1. With current or past medical history diseases or dysfunction that affect the clinical trial, evaluated by the investigator, including but not limited to central nervous system, cardiovascular system, respiratory system, digestive system, urinary system, endocrine system, blood system, ophthalmology and other diseases, history of malignant tumor or other diseases that are not suitable for participating in the clinical trial;
2. With current or previous mental disorders and brain dysfunction, or suicide risk according to the clinical judgment of the investigator, or a history of self-mutilation;
3. With any surgical condition or condition that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects participating in the trial, such as history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcers, history of gastrointestinal bleeding, etc.
4. With a known history of allergy to investigating drug ingredients or similar drugs, a history of allergic diseases or allergic constitution;
5. Positive for hepatitis B virus surface antigen (HBsAg), or syphilis antibody (Anti-TP), or hepatitis C antibody (anti-HCV), or human immunodeficiency virus antigen/antibody combined detection (HIV-Ag/Ab);
6. With a history of surgery within 3 months before screening, or have not recovered from surgery, or have an expected surgical plan during the trial;
7. With a blood donation or blood loss ≥ 400 mL within 3 months before screening, or a blood donation or blood loss ≥ 200 mL within 1 month, or a history of blood product use within 3 months before screening;
8. Taking any prescription drugs, over-the-counter drugs, and any functional vitamins or herbal products within 2 weeks before screening;
9. Using any drugs that inhibit or induce hepatic drug metabolizing enzymes CYP3A4, CYP3A5, CYP2D6 (such as inducers - phenobarbital, rifampicin, carbamazepine, phenytoin sodium, glucocorticoids, etc.; inhibitors - ketoconazole, itraconazole, cimetidine, clarithromycin, verapamil, erythromycin, etc.) within 4 weeks (or 5 half-lives, whichever is longer) before screening;
10. Participating in any clinical trial and taking clinical trial drugs within 3 months before screening, or being participating in other clinical trials;
11. Smoke test positive or smoking more than 5 cigarettes per day or average intake of coffee or tea more than 5 cups per day (200 mL/cup) within 3 months before screening, or unable to stop users during the study;
12. With alcohol abuse within 1 year before screening, average weekly alcohol intake more than 14 standard units [1 unit = 360 mL beer (alcohol content 5%) or 45 mL spirits (alcohol content 40%) or 150 mL wine (alcohol content 12%)] or positive for alcohol breath test;
13. With a history of drug abuse within 1 year before screening, or positive for urine drug screening;
14. With a family history of sudden cardiac death (sudden death age less than 40 years);
15. With a resting pulse < 50 beats/min or ≥ 100 beats/min; resting systolic blood pressure < 85 mmHg or ≥ 140 mmHg; resting diastolic blood pressure < 50 mmHg or ≥ 90 mmHg; systolic blood pressure decreased by ≥ 20 mmHg and/or diastolic blood pressure decreased by ≥ 10 mmHg and/or accompanied by clinical symptoms within 3 minutes of standing;
16. Abnormal in 12-lead electrocardiogram (ECG), clinically significant judged by the investigator (e.g., QTcF> 450 ms in men and > 470 ms in women);
17. With the aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatinine (Cr), urea (Urea), serum prolactin levels beyond the upper limit of normal (ULN);
18. Having special requirements for food, unable to observe a unified diet or having dysphagia;
19. Rejecting abide by the following conditions during the trial: smoking, alcohol or caffeine-containing beverages are prohibited, and strenuous exercise is avoided;
20. Directly related to this clinical trial;
21. Other subjects that the investigator considers inappropriate for this trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 23 days after treatment in part Ⅰ;
  Incidence of Treatment-Emergent Adverse Events
Incidence of Treatment-Emergent Adverse Events | 56 days after treatment in part Ⅱ;
  Incidence of Treatment-Emergent Adverse Events
Cmax | 360 hours after dosing in part Ⅰ;
  maximum observed plasma concentration of VV119 and the main metabolites
Cmax | 480 hours after dosing in part Ⅱ;
  maximum observed plasma concentration of the main metabolites VV119-M2
area under the plasma concentration time curve from time zero to the last(AUC0-t) | 360 hours after dosing in part Ⅰ;
  area under the plasma concentration time curve from time zero to the last of VV119 and the main metabolites
area under the plasma concentration time curve from time zero to the last(AUC0-t) | 480 hours after dosing in part Ⅱ;
  area under the plasma concentration time curve from time zero to the last of the main metabolites VV119-M2
AUC0-∞ | 360 hours after dosing in part Ⅰ;
  area under the plasma concentration time curve from time zero to infinity of VV119 and the main metabolites
AUC0-∞ | 480 hours after dosing in part Ⅱ;
  area under the plasma concentration time curve from time zero to infinity of the main metabolites VV119-M2
Tmax | 360 hours after dosing in part Ⅰ;
  time at which Cmax occurs of VV119 and the main metabolites of VV119 and the main metabolites
Tmax | 480 hours after dosing in part Ⅱ;
  time at which Cmax occurs of VV119 and the main metabolites of the main metabolites VV119-M2
t1/2 | 360 hours after dosing in part Ⅰ;
  half life of elimination of VV119 and the main metabolites
t1/2 | 480 hours after dosing in part Ⅱ;
  half life of elimination of the main metabolites VV119-M2
Apparent Clearance Rate（CL/F） | 360 hours after dosing in part Ⅰ;
  apparent clearance of VV119 and the main metabolites
Apparent Clearance Rate（CL/F） | 480 hours after dosing in part Ⅱ;
  apparent clearance of the main metabolites VV119-M2
Vd/F | 360 hours after dosing in part Ⅰ;
  apparent volume of distribution during the terminal phase of VV119 and the main metabolites
Vd/F | 480 hours after dosing in part Ⅱ;
  apparent volume of distribution during the terminal phase of the main metabolites VV119-M2
Ke | 360 hours after dosing in part Ⅰ;
  elimination rate constant of VV119 and the main metabolites
Ke | 480 hours after dosing in part Ⅱ;
  elimination rate constant of the main metabolites VV119-M2
mean Resident Time from time zero to the last（MRT0-t） | 360 hours after dosing in part Ⅰ;
  mean Resident Time from time zero to the last of VV119 of VV119 and the main metabolites
mean Resident Time from time zero to the last（MRT0-t） | 480 hours after dosing in part Ⅱ;
  mean Resident Time from time zero to the last of the main metabolites VV119-M2
mean Resident Time from time zero to infinity（MRT0-∞) | 360 hours after dosing in part Ⅰ;
  mean Resident Time from time zero to infinity of VV119 and the main metabolites
mean Resident Time from time zero to infinity（MRT0-∞) | 480 hours after dosing in part Ⅱ;
  mean Resident Time from time zero to infinity of the main metabolites VV119-M2
AUC_%Extra | 360 hours after dosing in part Ⅰ;
  area under plasma Concentration (AUC) extrapolated of VV119 and the main metabolites
AUC_%Extra | 480 hours after dosing in part Ⅱ;
  area under plasma Concentration (AUC) extrapolated of the main metabolites VV119-M2
BP | 360 hours after dosing in part Ⅰ;
  Blood Plasma Ratio of the main metabolites VV119-M2
BP | 480 hours after dosing in part Ⅱ;
  Blood Plasma Ratio of VV119 and the main metabolites

SECONDARY OUTCOMES:
Metabolite Identification | 360 hours after dosing
  Identification of the structure of the main metabolites of VV119 in plasma,Urine and feces

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Principal Investigator — Beijing Anding Hospital of Capital Medical University
Locations (1):
- Beijing Anding Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No